CLINICAL TRIAL: NCT02412787
Title: An Open Label Extension of Study HGT-HIT-094 Evaluating Long Term Safety and Clinical Outcomes of Intrathecal Idursulfase Administered in Conjunction With Elaprase® in Patients With Hunter Syndrome and Cognitive Impairment
Brief Title: Study of Long Term Safety and Clinical Outcomes of Idursulfase IT and Elaprase Treatment in Pediatric Participants Who Have Completed Study HGT-HIT-094
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP609-302; 2014-004143-13 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis II | interventions — idursulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idursulfase-IT (Experimental): Participants received 10 milligrams (mg) of idursulfase-IT intrathecally via intrathecal drug delivery device (IDDD) or lumbar puncture (LP) once every 28 days along with standard-of-care therapy with Elaprase, for 470 weeks (for participants who began intrathecal [IT] treatment in this study) and 480 weeks (for participants who began IT treatment in HGT-HIT-094 and continued to receive IT treatment in this study). Participants who were younger than 3 years of age received an adjusted dose of 7.5 mg (>8 months to 30 months of age) or 10 mg (>30 months to 3years of age) of idursulfase-IT.
  Interventions: Drug: Idursulfase-IT; Drug: Elaprase

INTERVENTIONS:
Drug: Idursulfase-IT — Participants received 10 mg of idursulfase-IT intrathecally via IDDD or LP once every 28 days. Participants who were younger than 3 years of age received an adjusted dose of 7.5 mg (>8 months to 30 months of age) and 10 mg (>30 months to 3 years of age).
  Other Names: HGT-2310
Drug: Elaprase — Participants received intravenous (IV) Elaprase infusions at a minimum of 48 hours after IT administration of idursulfase-IT.

SUMMARY:
This extension study will allow participants that completed Study HGT-HIT-094 to continue receiving Elaprase treatment in conjunction with idursulfase IT or to continue receiving Elaprase treatment and begin concurrent IT treatment for those that did not receive idursulfase IT treatment in Study HGT-HIT-094.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed Visit Week 52 assessments in Study HGT-HIT-094 (NCT02055118).
* The participant's parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form after all relevant aspects of the study have been explained and discussed. Consent of the participant's parent(s) or legally authorized guardian(s) and the participant's consent/assent, as relevant, must be obtained.
* The participant has continued to receive Elaprase on a regular basis in Study HGT-HIT-094 (NCT02055118).

Exclusion Criteria:

* The participant has experienced, in the opinion of the investigator, a safety or medical issue that contraindicates treatment with idursulfase-IT, including, but not limited to, uncontrolled seizure disorder, bleeding disorder, and clinically relevant hypertension.
* The participant has a known hypersensitivity to any of the components of idursulfase-IT.
* The participant has clinically relevant intracranial hypertension.
* The participant is enrolled in another clinical study, other than HGT-HIT-094 (NCT02055118), that involves clinical investigations or use of any investigational product (drug or [intrathecal/spinal] device) within 30 days prior to study enrollment or at any time during the study.
* The participant has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to compromised airways or other conditions.
* The participant has a condition that is contraindicated as described in the SOPH-A-PORT® Mini S, Implantable Access Port, Spinal, Mini Unattached, with Guidewire (SOPH-A-PORT Mini S) intrathecal drug delivery device (IDDD) Instructions for Use, including:

  1. The participant has had, or may have, an allergic reaction to the materials of construction of the SOPH-A-PORT Mini S device.
  2. The participant's body size is too small to support the size of the SOPH-A-PORT Mini S Access Port, as judged by the investigator.
  3. The participant's drug therapy requires substances known to be incompatible with the materials of construction.
  4. The participant has a known or suspected local or general infection.
  5. The participant is at risk of abnormal bleeding due to a medical condition or therapy.
  6. The participant has 1 or more spinal abnormalities that could complicate safe implantation or fixation.
  7. The participant has a functioning CSF shunt device.
  8. The participant has shown an intolerance to an implanted device.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (9):
- United States (3):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
- Women's and Children's Hospital, Adelaide, Australia
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Hôpital Femme Mère Enfants, Bron, France
- Instituto Nacional de Pediatría, Coyoacán, Mexico City, Mexico
- Hospital Infantil Universitario Niño Jesus, Madrid, Spain
- Royal Manchester Children's Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Yee KS, Chirila C, Davenport E, Mladsi D, Barnett C, Kronenberger WG. A post hoc analysis of Projected Retained Ability Scores (PRAS) for the longitudinal assessment of cognitive functioning in patients with neuronopathic mucopolysaccharidosis II receiving intrathecal idursulfase-IT. Orphanet J Rare Dis. 2023 Nov 2;18(1):343. doi: 10.1186/s13023-023-02957-2. PMID 37915038
- [Derived] Muenzer J, Burton BK, Harmatz P, Gutierrez-Solana LG, Ruiz-Garcia M, Jones SA, Guffon N, Inbar-Feigenberg M, Bratkovic D, Hale M, Wu Y, Yee KS, Whiteman DAH, Alexanderian D; SHP609-302 study group. Long-term open-label extension study of the safety and efficacy of intrathecal idursulfase-IT in patients with neuronopathic mucopolysaccharidosis II. Mol Genet Metab. 2022 Sep-Oct;137(1-2):92-103. doi: 10.1016/j.ymgme.2022.07.016. Epub 2022 Aug 2. PMID 35961250
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd54db2bf003ab46df0

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites in Australia, Canada, France, Mexico, Spain, the United Kingdom, and the United States of America (USA) from 14 April 2015 to 18 April 2024.
Pre-assignment Details: Participants who completed end of study (EOS) Visit Week 52 assessments of Study HGT-HIT-094 (NCT02055118) and who met the eligibility criteria were enrolled in this extension study. Some of the enrolled participants who were treated with idursulfase-IT in Study HGT-HIT-094 were analyzed as per the reference timepoints of HGT-HIT-094 study for some evaluations. For others, the reference timepoints after enrollment to the extension study were considered.
Groups:
- Idursulfase-IT: Participants received 10 milligrams (mg) of idursulfase-IT intrathecally via intrathecal drug delivery device (IDDD) or lumbar puncture (LP) once every 28 days along with standard-of-care therapy with Elaprase, for 470 weeks (for participants who began intrathecal [IT] treatment in this study) and 480 weeks (for participants who began IT treatment in HGT-HIT-094 and continued to receive IT treatment in this study). Participants who were younger than 3 years of age received an adjusted dose of 7.5 mg (>8 months to 30 months of age) or 10 mg (>30 months to 3 years of age) of idursulfase-IT.
Period: Overall Study
Arm/Group | Idursulfase-IT
Started | 56
Completed | 23
Not Completed | 33
Not completed — Withdrawal by Subject | 9
Not completed — Participation Terminated by Investigator | 1
Not completed — Site Terminated by Sponsor | 21
Not completed — Technical Problems | 1
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all the participants in Study SHP609-302 who underwent IDDD implantation or received at least 1 dose of study drug (full or partial).
Groups:
- Idursulfase-IT: Participants received 10 mg of idursulfase-IT intrathecally via IDDD or LP once every 28 days along with standard-of-care therapy with Elaprase, for 470 weeks (for participants who began IT treatment in this study) and 480 weeks (for participants who began IT treatment in HGT-HIT-094 and continued to receive IT treatment in this study). Participants who were younger than 3 years of age received an adjusted dose of 7.5 mg (>8 months to 30 months of age) or 10 mg (>30 months to 3 years of age) of idursulfase-IT.
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.89 (2.117)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 41
  More than one race | 0
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered investigational product-related.
Time Frame: Up to 9 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Participants | 56

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Participants were assessed for clinically significant changes in vital signs like injection (IT) vital signs and regular vital signs (temperature, pulse, blood pressure [systolic and diastolic], oxygen saturation, and respiration rate).
Time Frame: Up to 9 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Participants were assessed for clinically significant changes in laboratory parameters such as chemistry, hematology, urinalysis and cerebrospinal fluid (CSF) values.
Time Frame: Up to 9 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Findings
Description: Participants were assessed for clinically significant changes in 12-lead ECG findings (such as heart rate, PR interval, QRS interval, QT interval, and the corrected QT interval).
Time Frame: Up to 9 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Participants | 0

5. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Idursulfase
Description: Idursulfase concentrations in serum were determined using a validated Enzyme -Linked Immunosorbent Assay (ELISA) method. Concentration for Cmax is presented in this endpoint.
Time Frame: Predose and at 30 min, 60 min, 120 min, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 30 hours and 36 hours post-dose at Week 100 in relation to HGT-HIT-094 (Week 48 of this study)
Population: The Pharmacokinetic Population included all the participants in Study SHP609-302 who received study drug and participated in the scheduled pharmacokinetic studies, and for whom at least 1 post-dose pharmacokinetic blood sample was collected. Overall number of participants analyzed is the number of participants with data available for analyses. Participants were divided into 3 groups for this outcome measure based on the time they received IT treatment in relation to prior study HGT-HIT-094.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Idursulfase-IT 10 mg, Delayed IT: The Delayed IT group included participants who were randomized to the no IT treatment cohort in Study HGT-HIT-094 and began IT treatment in Study SHP609-302.
- Idursulfase-IT 10 mg, Early IT: The Early IT group included participants who were randomized to the IT treatment cohort in Study HGT-HIT-094 and continued in Study SHP609-302.
- Idursulfase-IT 10 mg, Former Substudy: The Former Substudy group included participants who received IT treatment in HGT-HIT-094 substudy.
Arm/Group | Idursulfase-IT 10 mg, Delayed IT | Idursulfase-IT 10 mg, Early IT | Idursulfase-IT 10 mg, Former Substudy
Number analyzed (Participants) | 10 | 20 | 3
nanograms per milliliter (ng/mL) | 128.19 (169.427) | 104.89 (66.879) | 120.23 (57.308)

6. Other Pre Specified Outcome: Maximum Observed Concentration (Cmax) of Idursulfase in Cerebrospinal Fluid (CSF)
Description: Data was not collected for this outcome measure due to Sponsor decision.
Time Frame: Predose each week up to 9 years
Reporting Status: Not Posted

7. Primary Outcome: Percent Change From Baseline in the Concentration of Glycosaminoglycan (GAG) in CSF at Month 67
Description: The percent change in concentration of GAG in CSF was assessed. GAGs are long sugar chains that are like building blocks for the body's tissues, especially connective tissues like cartilage, skin, and tendons, and play a crucial role in cell signaling and interactions.
Time Frame: For participants who began IT treatment in HGT-HIT-094: From Baseline of HGT-HIT-094 up to Month 67 in relation to HGT-HIT-094; For participants who began IT treatment in this study: From Baseline of this study up to Month 55 of this study.
Population: The Safety Population included all the participants in Study SHP609-302 who underwent IDDD implantation or received at least 1 dose of study drug (full or partial). Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 27
percent change | -71.15 (17.842)

8. Primary Outcome: Percent Change From Baseline in the Concentration of GAG in Urine at Month 67
Description: The percent change in concentration of GAG in urine was assessed. GAGs are long sugar chains that are like building blocks for the body's tissues, especially connective tissues like cartilage, skin, and tendons, and play a crucial role in cell signaling and interactions.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 23
percent change | -32.44 (29.366)

9. Primary Outcome: Number of Participants Who Reported Positive for Anti-idursulfase Antibodies in CSF
Time Frame: Up to 9 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Participants | 25

10. Primary Outcome: Number of Participants Who Reported Positive for Anti-idursulfase Antibodies in Serum
Time Frame: Up to 9 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 56
Participants | 46

11. Secondary Outcome: Change From Baseline in Differential Ability Scales, Second Edition (DAS-II) Standard Cluster Scores at Month 67
Description: DAS-II was used to assess all participants of age 2 years, 6 months or older. DAS-II comprises 2 overlapping batteries. Early Years battery (EYB) was designed for children ages 2 years, 6 months through 6 years, 11 months. The School Age Battery (SAB) was designed for children ages 7 years, 0 months through 17 years, 11months. These batteries are fully co-normed for ages 5 years, 0 months, through 8 years, 11 months. The cluster areas include general conceptual ability (GCA), verbal, nonverbal, spatial, and special nonverbal composite (SNC). The cluster area score represents a score (mean=100 and standard deviation=15) on which higher scores indicate higher level of cognitive ability.
Time Frame: as for outcome 7
Population: The Safety Population included all the participants in Study SHP609-302 who underwent IDDD implantation or received at least 1 dose of study drug (full or partial). Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants available for analyses for the specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 3
score on a scale
  GCA: number analyzed (Participants) | 2
  GCA | -6.0 (8.49)
  Verbal | -23.7 (21.59)
  Nonverbal: number analyzed (Participants) | 2
  Nonverbal | -20.5 (7.78)
  Spatial | 0.3 (18.88)
  SNC: number analyzed (Participants) | 2
  SNC | -5.5 (6.36)

12. Other Pre Specified Outcome: Change From Baseline in Age Equivalent Scores of the Bayley Scales of Infant Development, Third Edition (BSID-III) Domains
Description: This pre-specified optional outcome measure was not assessed.
Time Frame: as for outcome 7
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change From Baseline in Development Quotient (DQ) of the Bayley Scales of Infant Development, Third Edition (BSID-III) Domains
Description: This pre-specified optional outcome measure was not assessed.
Time Frame: as for outcome 7
Reporting Status: Not Posted

14. Secondary Outcome: Change From Baseline in Standard Scores of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) Domains at Month 67
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite [ABC] (a composite of the other 4 domains). The standard scores for four key domains were mean=100 and standard deviation=15, where higher scores indicate a higher level of cognitive ability. Positive change from baseline indicates improvement in adaptive functioning. The ABC score (a composite of the other 4 domains) ranges from 20 to 160 on which higher scores indicate a higher level of adaptive functioning. A positive change from baseline value indicates improvement in adaptive functioning.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  Communication | -13.5 (4.95)
  Daily Living Skills | -9.5 (0.71)
  Socialization | -14.5 (9.19)
  Motor Skills | 11.5 (7.78)
  ABC | -13.5 (2.12)

15. Secondary Outcome: Change From Baseline in Standard Composite Scores of the VABS-II Domains at Month 67
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the ABC (a composite of the other 4 domains). The ABC score ranges from 20 to 160 on which higher scores indicate a higher level of adaptive functioning. A positive change value indicates improvement in adaptive functioning.
Time Frame: as for outcome 7
Population: The Safety Population included all the participants in Study SHP609-302 who underwent IDDD implantation or received at least 1 dose of study drug (full or partial). Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for the specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  Baseline Age <6 Years | -13.5 (2.12)
  Baseline Age ≥6 Years: number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline in Age Equivalents Score of the Differential Ability Scales, Second Edition (DAS-II) at Month 61
Description: DAS-II comprises 2 overlapping batteries; EYB= 2 years,6 months through 6 years,11 months and SAB=7 years,0 months through 17 years,11 months. Core subtests include Verbal Comprehension, Picture Similarities, Naming Vocabulary, Pattern Construction, Matrices and Copying for DAS-II Early Years and Recall of Designs, Word Definitions, Pattern Construction, Matrices, Verbal Similarities, and Sequential and Quantitative Reasoning for DAS-II School Years. Standard subtests scores (mean=50 and standard deviation of 10) for each subtest were converted to age equivalent scores (AES). Higher AES indicates greater cognitive ability. Negative change from baseline indicates worsening.
Time Frame: For participants who began IT treatment in HGT-HIT-094: From Baseline of HGT-HIT-094 up to Month 61 in relation to HGT-HIT-094; For participants who began IT treatment in this study: From Baseline of this study up to Month 49 of this study.
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  EYB: Verbal Comprehension | 1.50 (1.768)
  EYB: Picture Similarities | 2.63 (2.652)
  EYB: Naming Vocabulary | 3.13 (1.237)
  EYB: Pattern Construction | 1.38 (1.237)
  EYB: Matrices | 3.38 (1.237)
  EYB: Copying | 1.13 (1.591)
  SAB: Recall of Designs: number analyzed (Participants) | 1
  SAB: Recall of Designs | 0.00 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Word Definitions: number analyzed (Participants) | 1
  SAB: Word Definitions | -0.25 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Pattern Construction: number analyzed (Participants) | 1
  SAB: Pattern Construction | 0.00 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Matrices: number analyzed (Participants) | 1
  SAB: Matrices | 2.50 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Verbal Similarities: number analyzed (Participants) | 1
  SAB: Verbal Similarities | 0.00 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Sequential & Quantitative Reasoning: number analyzed (Participants) | 1
  SAB: Sequential & Quantitative Reasoning | 0.75 (NA) — Standard deviation was not estimable for a single participant.

17. Secondary Outcome: Change From Baseline in Developmental Quotients (DQ) of the DAS-II at Month 61
Description: DAS-II was used to assess all participants of age 2 years,6 months or older.DAS-II comprises 2 overlapping batteries.EYB was designed for children ages 2 years,6 months through 6 years,11 months.SAB was designed for children ages 7 years,0 months through 17 years,11 months.Core subtests include Verbal Comprehension,Picture Similarities,Naming Vocabulary,Pattern Construction,Matrices, & Copying for DAS-II Early Years&Recall of Designs,Word Definitions, Pattern Construction,Matrices,Verbal Similarities, & Sequential and Quantitative Reasoning for the DAS-II School Years. The DQ was computed as a ratio and expressed as a percentage using the AES divided by the age at testing ([AES/chronological age] × 100; range, 0-100). The higher score indicates greater cognitive ability. The subtest score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability. A positive change value indicates improvement in cognitive ability.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  EYB: Verbal Comprehension | -27.45 (13.223)
  EYB: Picture Similarities | -7.75 (23.971)
  EYB: Naming Vocabulary | -10.95 (4.596)
  EYB: Pattern Construction | -22.25 (7.425)
  EYB: Matrices | -9.20 (12.021)
  EYB: Copying | -34.95 (15.627)
  SAB: Recall of Designs: number analyzed (Participants) | 1
  SAB: Recall of Designs | -25.90 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Word Definitions: number analyzed (Participants) | 1
  SAB: Word Definitions | -29.30 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Pattern Construction: number analyzed (Participants) | 1
  SAB: Pattern Construction | -28.50 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Matrices: number analyzed (Participants) | 1
  SAB: Matrices | 2.20 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Verbal Similarities: number analyzed (Participants) | 1
  SAB: Verbal Similarities | -25.90 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Sequential & Quantitative Reasoning: number analyzed (Participants) | 1
  SAB: Sequential & Quantitative Reasoning | -19.80 (NA) — Standard deviation was not estimable for a single participant.

18. Secondary Outcome: Change From Baseline in T-scores of the Core Subtests DAS-II at Month 61
Description: DAS-II was used to assess all participants of age 2 years, 6 months or older. DAS-II comprises 2 overlapping batteries. EYB was designed for children ages 2 years, 6 months through 6 years, 11 months. SAB was designed for children ages 7 years, 0 months through 17 years, 11months. The core subtests include Verbal Comprehension, Picture Similarities, Naming Vocabulary, Pattern Construction, Matrices, and Copying for the DAS-II Early Years and Recall of Designs, Word Definitions, Pattern Construction, Matrices, Verbal Similarities, and Sequential and Quantitative Reasoning for the DAS-II School Years. Core subtests score represent a score (mean = 50 and standard deviation of 10) on which higher scores indicate a higher level of cognitive ability.
Time Frame: as for outcome 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  EYB: Verbal Comprehension | -14.5 (9.19)
  EYB: Picture Similarities | -6.5 (10.61)
  EYB: Naming Vocabulary | -8.5 (4.95)
  EYB: Pattern Construction | -10.0 (9.90)
  EYB: Matrices | 2.5 (2.12)
  EYB: Copying | -14.0 (26.87)
  SAB: Recall of Designs: number analyzed (Participants) | 1
  SAB: Recall of Designs | -4.0 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Word Definitions: number analyzed (Participants) | 1
  SAB: Word Definitions | -28.0 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Pattern Construction: number analyzed (Participants) | 1
  SAB: Pattern Construction | -13.0 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Matrices: number analyzed (Participants) | 1
  SAB: Matrices | -3.0 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Verbal Similarities: number analyzed (Participants) | 1
  SAB: Verbal Similarities | -24.0 (NA) — Standard deviation was not estimable for a single participant.
  SAB: Sequential & Quantitative Reasoning: number analyzed (Participants) | 1
  SAB: Sequential & Quantitative Reasoning | -2.0 (NA) — Standard deviation was not estimable for a single participant.

19. Secondary Outcome: Change From Baseline in Age Equivalents Score of the VABS-II Sub Domains at Month 67
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following subdomains of 5 key domains: Communication (Receptive, Expressive, Written), Daily Living Skills(Personal, Domestic, Community), Socialization (Interpersonal Relationships, Play and Leisure Time, Coping Skills), Motor Skills (Gross, Fine). Standard subdomain scores (mean=100 and standard deviation of 15) for each subdomain were converted to AES. Higher AES indicates greater cognitive ability. Negative change from baseline indicates worsening.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  Communication: Receptive | 2.13 (0.412)
  Communication: Expressive | 2.54 (1.591)
  Communication: Written | 1.58 (1.296)
  Daily Living Skills: Personal | 4.50 (1.296)
  Daily Living Skills: Domestic | 3.42 (0.825)
  Daily Living Skills: Community | 1.83 (0.943)
  Socialization: Interpersonal Relationships | 1.92 (4.832)
  Socialization: Play and Leisure Time | 2.25 (1.768)
  Socialization: Coping Skills | 0.75 (1.296)
  Motor Skills: Gross | 9.75 (8.721)
  Motor Skills: Fine | 2.33 (0.118)

20. Secondary Outcome: Change From Baseline in DQ of the VABS-II Sub Domains at Month 67
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following subdomains of 5 key domains: Communication (Receptive, Expressive, Written), Daily Living Skills (Personal, Domestic, Community), Socialization (Interpersonal Relationships, Play and Leisure Time, Coping Skills), Motor Skills (Gross, Fine). The DQ was computed as a ratio and expressed as a percentage using the age-equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range, 0-100). Higher scores indicate better cognitive ability. A positive change from baseline value indicates improvement in cognition.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  Communication: Receptive | -7.30 (19.375)
  Communication: Expressive | -6.65 (23.547)
  Communication: Written | -40.15 (10.677)
  Daily Living Skills: Personal | 9.50 (13.011)
  Daily Living Skills: Domestic | -22.60 (0.424)
  Daily Living Skills: Community | -27.15 (16.900)
  Socialization: Interpersonal Relationships | -26.00 (44.265)
  Socialization: Play and Leisure Time | -18.00 (13.435)
  Socialization: Coping Skills | -44.65 (31.183)
  Motor Skills: Gross | 47.35 (66.539)
  Motor Skills: Fine | -19.90 (6.788)

21. Secondary Outcome: Change From Baseline in v-Scores of the VABS-II Sub Domains at Month 67
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following subdomains of 5 key domains: Communication (Receptive, Expressive, Written), Daily Living Skills (Personal, Domestic, Community), Socialization (Interpersonal Relationships, Play and Leisure Time, Coping Skills), Motor Skills (Gross, Fine). The V-scale scores represent a score (mean = 15 and standard deviation of 3; range: 1-24) on which higher scores indicate a higher level of adaptive functioning.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 2
score on a scale
  Communication: Receptive | -0.5 (2.12)
  Communication: Expressive | -1.0 (2.83)
  Communication: Written | -8.0 (2.83)
  Daily Living Skills: Personal | 1.0 (1.41)
  Daily Living Skills: Domestic | -2.0 (1.41)
  Daily Living Skills: Community | -5.0 (1.41)
  Socialization: Interpersonal Relationships | -3.0 (5.66)
  Socialization: Play and Leisure Time | -2.0 (1.41)
  Socialization: Coping Skills | -3.5 (2.12)
  Motor Skills: Gross | 2.5 (2.12)
  Motor Skills: Fine | 1.5 (0.71)

22. Secondary Outcome: Change From Baseline in v-Scale Scores of the VABS-II Maladaptive Behavior Index and Its Subscales at Month 67
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. The maladaptive behavior index is a composite of the internalizing, externalizing, and other types of undesirable behavior that may interfere with the individual's adaptive functioning. The v-Scale scores represent a score (mean = 15 and standard deviation of 3; range: 1-24) on which higher scores indicate a higher level of adaptive functioning.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 1
score on a scale
  Maladaptive Behavior Index | -3.0 (NA) — Standard deviation was not estimable for a single participant.
  Internalizing | -4.0 (NA) — Standard deviation was not estimable for a single participant.
  Externalizing | -1.0 (NA) — Standard deviation was not estimable for a single participant.

23. Secondary Outcome: Number of Participants With Observed Maladaptive Levels of the VABS-II Maladaptive Behavior Index and Its Subscales at Month 61
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. The maladaptive behavior index is a composite of the internalizing, externalizing, and other types of undesirable behavior that may interfere with the individual's adaptive functioning. Only categories having non-zero values are reported.
Time Frame: For participants who began IT treatment in HGT-HIT-094: At Month 61 in relation to HGT-HIT-094; For participants who began IT treatment in this study: At Month 49 of this study.
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 47
Participants
  Maladaptive Behavior Index; Average | 7
  Maladaptive Behavior Index; Elevated | 1
  Internalizing; Average | 6
  Internalizing; Elevated | 2
  Externalizing; Average | 2
  Externalizing; Elevated | 6

24. Secondary Outcome: Change From Baseline in Brain Structure Volume as Measured by Magnetic Resonance Imaging (MRI)
Description: Brain structure volume was assessed from brain total intracranial volume, brain total tissue volume, brain total white matter, brain total gray matter, and total CSF volume as measured by MRI.
Time Frame: For participants who began IT treatment in HGT-HIT-094: From Baseline of HGT-HIT-094 up to Month 120 in relation to HGT-HIT-094; For participants who began IT treatment in this study: From Baseline of this study up to Month 108 of this study.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cubic centimeters (cm^3)
Arm/Group | Idursulfase-IT
Number analyzed (Participants) | 3
cubic centimeters (cm^3)
  Brain Total Intracranial Volume | -19.813 (70.994)
  Brain Total Tissue Volume | -38.573 (134.021)
  Brain Total White Matter Volume | 98.180 (64.194)
  Brain Total Gray Matter Volume | -136.750 (79.547)
  Total CSF Volume | 58.480 (52.382)

ADVERSE EVENTS:
Time Frame: Up to 9 years
Description: The Safety Population included all the participants in Study SHP609-302 who underwent IDDD implantation or received at least 1 dose of study drug (full or partial).
Arm/Group | Idursulfase-IT
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 48/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idursulfase-IT (N=56)
Abdominal pain (Gastrointestinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Albumin CSF increased (Investigations) | 1
Anaphylactic reaction (Immune system disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bacteraemia (Infections and infestations) | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
CSF cell count increased (Investigations) | 1
CSF glucose decreased (Investigations) | 1
CSF lymphocyte count increased (Investigations) | 1
CSF protein increased (Investigations) | 1
CSF white blood cell count (Investigations) | 1
Campylobacter infection (Infections and infestations) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Catheter site cellulitis (Infections and infestations) | 1
Central nervous system infection (Infections and infestations) | 3
Cerebrospinal fluid leakage (Nervous system disorders) | 12
Cholelithiasis (Hepatobiliary disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Convulsion (Nervous system disorders) | 2
Corona virus infection (Infections and infestations) | 2
Deafness (Ear and labyrinth disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Device breakage (General disorders) | 4
Device deployment issue (General disorders) | 1
Device dislocation (General disorders) | 3
Device extrusion (General disorders) | 1
Device failure (General disorders) | 22
Device kink (General disorders) | 4
Device malfunction (General disorders) | 1
Device misuse (General disorders) | 1
Device related infection (Infections and infestations) | 4
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1
Endocarditis (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 1
Gastroenteritis viral (Infections and infestations) | 1
Haematochezia (Gastrointestinal disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hyperthermia (General disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothermia (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Implant site abscess (Infections and infestations) | 1
Implant site effusion (General disorders) | 1
Implant site infection (Infections and infestations) | 1
Inflammation (General disorders) | 1
Influenza (Infections and infestations) | 3
Injection site swelling (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Medical device site reaction (General disorders) | 1
Meningitis bacterial (Infections and infestations) | 2
Meningitis streptococcal (Infections and infestations) | 1
Nocardiosis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Pleocytosis (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 2
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Procedural vomiting (Injury, poisoning and procedural complications) | 2
Pseudomeningocele (Injury, poisoning and procedural complications) | 2
Pyrexia (General disorders) | 10
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory syncytial virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sleep disorder (Psychiatric disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Staphylococcus test positive (Investigations) | 1
Staring (Psychiatric disorders) | 1
Stenotrophomonas infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Testicular torsion (Reproductive system and breast disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tonsillitis (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 1
Vascular complication associated with device (General disorders) | 7
Vomiting (Gastrointestinal disorders) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idursulfase-IT (N=56)
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 4
Abnormal behaviour (Psychiatric disorders) | 8
Achilles tendon discomfort (Musculoskeletal and connective tissue disorders) | 3
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 4
Adenovirus infection (Infections and infestations) | 3
Aggression (Psychiatric disorders) | 11
Agitation (Psychiatric disorders) | 8
Alanine aminotransferase increased (Investigations) | 11
Albumin CSF increased (Investigations) | 12
Anaemia (Blood and lymphatic system disorders) | 5
Anxiety (Psychiatric disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthropod bite (Injury, poisoning and procedural complications) | 10
Aspartate aminotransferase increased (Investigations) | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Astigmatism (Eye disorders) | 4
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 16
Blister (Skin and subcutaneous tissue disorders) | 3
Blood bicarbonate decreased (Investigations) | 8
Blood calcium decreased (Investigations) | 3
Blood pressure diastolic decreased (Investigations) | 12
Blood pressure diastolic increased (Investigations) | 13
Blood pressure increased (Investigations) | 6
Blood pressure systolic decreased (Investigations) | 14
Blood pressure systolic increased (Investigations) | 14
Blood thyroid stimulating hormone increased (Investigations) | 5
Blood triglycerides increased (Investigations) | 13
Blood uric acid increased (Investigations) | 3
Body temperature decreased (Investigations) | 12
Bronchitis (Infections and infestations) | 5
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
CSF cell count increased (Investigations) | 13
CSF glucose decreased (Investigations) | 16
CSF neutrophil count increased (Investigations) | 3
CSF protein increased (Investigations) | 20
CSF test abnormal (Investigations) | 4
CSF white blood cell count increased (Investigations) | 12
Carbon dioxide decreased (Investigations) | 9
Cardiac murmur (Investigations) | 3
Carpal tunnel syndrome (Nervous system disorders) | 16
Catheter site effusion (General disorders) | 6
Catheter site erythema (General disorders) | 6
Catheter site extravasation (General disorders) | 5
Catheter site pain (General disorders) | 3
Catheter site swelling (General disorders) | 6
Cerebrospinal fluid retention (Nervous system disorders) | 3
Cerumen impaction (Ear and labyrinth disorders) | 3
Choking (Respiratory, thoracic and mediastinal disorders) | 3
Conjunctivitis (Eye disorders) | 8
Constipation (Gastrointestinal disorders) | 12
Contusion (Injury, poisoning and procedural complications) | 12
Corona virus infection (Infections and infestations) | 17
Coronavirus test positive (Investigations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 40
Croup infectious (Infections and infestations) | 3
Deafness (Ear and labyrinth disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 10
Dental caries (Gastrointestinal disorders) | 15
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 10
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 3
Device breakage (General disorders) | 6
Device malfunction (General disorders) | 17
Device occlusion (General disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 30
Diastolic hypertension (Vascular disorders) | 5
Diastolic hypotension (Vascular disorders) | 5
Drug hypersensitivity (Immune system disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Dysphemia (Psychiatric disorders) | 3
Ear infection (Infections and infestations) | 32
Ear pain (Ear and labyrinth disorders) | 8
Eczema (Skin and subcutaneous tissue disorders) | 4
Electrocardiogram QT prolonged (Investigations) | 5
Enuresis (Renal and urinary disorders) | 4
Eosinophil count increased (Investigations) | 12
Eosinophil percentage increased (Investigations) | 6
Eosinophilia (Blood and lymphatic system disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 9
Excoriation (Injury, poisoning and procedural complications) | 14
Eye swelling (Eye disorders) | 5
Face oedema (General disorders) | 4
Fall (Injury, poisoning and procedural complications) | 17
Fatigue (General disorders) | 6
Febrile convulsion (Nervous system disorders) | 3
Flushing (Vascular disorders) | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 6
Foramen magnum stenosis (Congenital, familial and genetic disorders) | 3
Frequent bowel movements (Gastrointestinal disorders) | 3
Fungal skin infection (Infections and infestations) | 3
Gait disturbance (General disorders) | 13
Gastroenteritis (Infections and infestations) | 11
Gastroenteritis viral (Infections and infestations) | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Haematochezia (Gastrointestinal disorders) | 3
Haematocrit decreased (Investigations) | 8
Haemoglobin decreased (Investigations) | 9
Hand-foot-and-mouth disease (Infections and infestations) | 3
Head injury (Injury, poisoning and procedural complications) | 4
Headache (Nervous system disorders) | 27
Heart rate decreased (Investigations) | 15
Heart rate increased (Investigations) | 15
Hepatomegaly (Hepatobiliary disorders) | 3
Hypersensitivity (Immune system disorders) | 3
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 6
Implant site effusion (General disorders) | 7
Implant site swelling (General disorders) | 3
Incision site oedema (Injury, poisoning and procedural complications) | 10
Incision site pain (Injury, poisoning and procedural complications) | 4
Influenza (Infections and infestations) | 18
Influenza like illness (General disorders) | 3
Infusion site swelling (General disorders) | 3
Insomnia (Psychiatric disorders) | 7
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Iron deficiency (Metabolism and nutrition disorders) | 6
Irritability (General disorders) | 11
Joint injury (Injury, poisoning and procedural complications) | 4
Laceration (Injury, poisoning and procedural complications) | 9
Laryngitis (Infections and infestations) | 3
Lethargy (Nervous system disorders) | 7
Ligament sprain (Injury, poisoning and procedural complications) | 5
Lower respiratory tract infection (Infections and infestations) | 3
Medical device complication (General disorders) | 9
Medical device pain (General disorders) | 4
Metapneumovirus infection (Infections and infestations) | 3
Middle ear effusion (Ear and labyrinth disorders) | 4
Motion sickness (Ear and labyrinth disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24
Nasopharyngitis (Infections and infestations) | 38
Nausea (Gastrointestinal disorders) | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Nerve compression (Nervous system disorders) | 3
Neutrophil count decreased (Investigations) | 3
Neutrophil count increased (Investigations) | 8
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 6
Ocular hyperaemia (Eye disorders) | 3
Oral herpes (Infections and infestations) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Otitis externa (Infections and infestations) | 6
Otitis media (Infections and infestations) | 21
Otitis media acute (Infections and infestations) | 12
Otorrhoea (Ear and labyrinth disorders) | 12
Oxygen saturation decreased (Investigations) | 11
Pain (General disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17
Pharyngitis (Infections and infestations) | 5
Pharyngitis streptococcal (Infections and infestations) | 10
Platelet count decreased (Investigations) | 7
Pneumonia (Infections and infestations) | 7
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3
Procedural headache (Injury, poisoning and procedural complications) | 5
Procedural hypertension (Injury, poisoning and procedural complications) | 9
Procedural hypotension (Injury, poisoning and procedural complications) | 13
Procedural nausea (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 33
Procedural vomiting (Injury, poisoning and procedural complications) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Proteinuria (Renal and urinary disorders) | 3
Pseudomeningocele (Injury, poisoning and procedural complications) | 5
Psychomotor hyperactivity (Nervous system disorders) | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Pyrexia (General disorders) | 43
Rash (Skin and subcutaneous tissue disorders) | 16
Rash erythematous (Skin and subcutaneous tissue disorders) | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Red blood cell count decreased (Investigations) | 9
Red blood cells CSF positive (Investigations) | 7
Red man syndrome (Skin and subcutaneous tissue disorders) | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory syncytial virus infection (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 5
Retching (Gastrointestinal disorders) | 3
Rhinitis (Infections and infestations) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 25
Scab (Skin and subcutaneous tissue disorders) | 4
Scoliosis (Musculoskeletal and connective tissue disorders) | 3
Scratch (Injury, poisoning and procedural complications) | 5
Seasonal allergy (Immune system disorders) | 7
Sinus bradycardia (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 8
Sinusitis (Infections and infestations) | 11
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5
Sleep disorder (Psychiatric disorders) | 7
Spinal disorder (Musculoskeletal and connective tissue disorders) | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3
Staphylococcal infection (Infections and infestations) | 3
Staring (Psychiatric disorders) | 5
Swelling face (Skin and subcutaneous tissue disorders) | 4
Systolic hypertension (Vascular disorders) | 4
Tachycardia (Cardiac disorders) | 4
Thermal burn (Injury, poisoning and procedural complications) | 3
Tinea pedis (Infections and infestations) | 4
Toe walking (Musculoskeletal and connective tissue disorders) | 7
Tooth abscess (Infections and infestations) | 4
Tooth fracture (Injury, poisoning and procedural complications) | 4
Tooth infection (Infections and infestations) | 8
Toothache (Gastrointestinal disorders) | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 3
Umbilical hernia (Gastrointestinal disorders) | 4
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 37
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Urinary tract infection (Infections and infestations) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 10
Vascular complication associated with device (General disorders) | 9
Viral infection (Infections and infestations) | 8
Vomiting (Gastrointestinal disorders) | 40
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9
White blood cell count decreased (Investigations) | 4
White blood cell count increased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT02412787/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT02412787/SAP_001.pdf